CLINICAL TRIAL: NCT05833412
Title: Clinical Study to Improve the Quality of Care in Critically Ill Patients With Suspected Sepsis Through Early Molecular Diagnosis .
Brief Title: Molecular Early Sepsis Identification Study
Acronym: MESIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Alejandro Rodriguez Oviedo , MD (Other)
Collaborators: BioMérieux (Industry); Biocartis NV (Industry)
Responsible Party: Sponsor-Investigator, Alejandro Rodriguez Oviedo , MD, MD,PhD,MSc, Hospital Universitari Joan XXIII de Tarragona.
Organization: Hospital Universitari Joan XXIII de Tarragona. (Other)
Other Study IDs: 182/2022
Record Dates: First submitted 2023-04-17; First posted 2023-04-27 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Sepsis; Molecular Diagnosis
Keywords: sepsis; Molecular diagnosis; Filmarrays
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Suspected sepsis: These patients will undergo molecular diagnosis by performing the Septicyte Rapid® test on whole blood (EDTA) which allows to know the risk of sepsis (low, intermediate, high) and after 6-8 hours of blood culture incubation, filmarrays blood culture identification (BCID2®) a molecular test approved for direct identification of BSI causing pathogens from blood culture will be performed.
  Interventions: Diagnostic Test: Septicyte Rapid ®; Diagnostic Test: FilmArray® blood culture identification (BCID2®)

INTERVENTIONS:
Diagnostic Test: Septicyte Rapid ® — SeptiCyte RAPID is based on the measurement of two gene expression biomarkers in peripheral blood (PLAC8 and PLA2G7) using quantitative reverse transcription-polymerase chain reaction (RT-qPCR). Based on the results obtained in 1 hour from whole blood (100 mcl), the device issues a report with a sepsis probability scale according to 4 bands (1 low probability, 2-3 intermediate probability and 4 high probability).
Diagnostic Test: FilmArray® blood culture identification (BCID2®) — After 6 to 8 hours of blood culture incubation, BCID2 will be performed on each of the 4 bottles. The BCID2 assay is an approved molecular test for the direct identification of pathogens causing bloodstream infections from blood cultures. The BCID2 Panel analyzes 43 targets associated with bloodstream infections, including Gram-negative bacteria, Gram-positive bacteria, yeasts and 10 antimicrobial resistance genes, all with a single test and with results available in approximately one hour from the blood culture. In addition, the BCID2® Panel menu includes seven additional resistance genes, including carbapenemases, colistin resistance genes and a MREJ assay that enables more speciﬁc MRSA identiﬁcation.

SUMMARY:
Single-center, retrospective observational study to evaluate the implementation of early molecular diagnosis of sepsis using SeptiCyte and BCID2 in 120 critically ill patients with suspected sepsis without clear focus and requiring antimicrobial treatment.

The main objective is to evaluate the performance of these molecular techniques with respect to routine clinical practice and their impact on the optimization of antimicrobial treatment in this group of patients.

DETAILED DESCRIPTION:
Background Sepsis has recently been redefined (Sepsis 3) as an infection leading to organ dysfunction (1). Although this definition is not generally accepted by all researchers (2,3) due to the potential for delayed diagnosis, mortality related to this entity could be significantly reduced by early adoption of diagnostic protocols and appropriate and early use of antimicrobial therapy (ATB).

A recent study in Catalonia (4) showed an incidence of 212 cases of sepsis per 100,000 inhabitants/year with a hospital mortality of 21%, which is significantly higher if consider ICU patients (40%) or those affected by septic shock (>50%) (5,6). These data highlight the current importance of this entity and highlight the need to seek new alternatives for early and appropriate diagnosis and treatment to have a favourable impact on the high mortality rate.

Ineffective treatment of sepsis is often due to late diagnosis of sepsis, due to the inherent complication of nonspecific clinical signs. Although procalcitonin (PCT) appears to be an adequate biomarker for the diagnosis of bacterial infection (7,8), different studies show a discrimination of only around 80% (7,8) and recent international guidelines do not recommend its use (9,10,11). These same guidelines recommend the use of scores, such as SOFA (sequential organ failure assessment) and qSOFA (a simplified version) based on the presence of altered consciousness, hypotension, and tachypnoea) for early risk stratification of patients suspected of infection.

However, sepsis and non-sepsis systemic inflammatory syndromes present as clinically similar entities, and both are frequently complicated by the appearance of organ dysfunction. Therefore, the identification of sepsis remains subjective and possibly leads to overdiagnosis of sepsis and consequently a high use of ATB in patients who do not have sepsis and who do not benefit from this treatment (12).

The availability of new molecular techniques and the automation of these laboratory analyses have stimulated the search for biomarkers related to the host response to sepsis. Analysis of host gene expression through RNA transcripts (transcriptomics) offers an opportunity in this complex setting of the critically ill patient. Host gene expression differs greatly between septic patients and healthy individuals (13). However, although gene expression between septic and non-septic inflamed patients overlaps to a large extent, several differences between transcripts observed in sepsis can help distinguish infection from other causes of inflammation [14]. The SeptiCyte™ LAB transcription assay was developed to diagnose infection in critically ill patients with suspected sepsis [15]. It is the first host response assay based on quantitative reverse transcriptase PCR (qRT-PCR) methods to be approved by the US Food and Drug Administration (FDA). SeptiCyte™ LAB allows the assessment of host response to infection by measuring the expression of specific genes involved in immune function and inflammatory signaling in whole blood. The first clinical performance study of SeptiCyte™ LAB analyzed 345 patients who were enrolled as part of the Molecular Diagnosis and Sepsis Risk Stratification (MARS) cohort in two ICUs in the Netherlands [15]. Patients were categorized as having sepsis based on a post-hoc medical assessment of the available clinical, radiological, and microbiological evidence [16] resulting in estimates for the AUC (0.77 to 0.99), sensitivity (79% to 100%) and specificity (33% to 91%) varied widely, depending on the prevalence of sepsis, the confidence level with respect to the reference diagnosis and whether patient registration was consecutive. As this analysis took about 6 hours, an early sepsis diagnostic tool (SeptiCyte RAPID (17) has been developed that is based on the measurement of two of the four gene expression biomarkers in peripheral blood (PLAC8 and PLA2G7) using the same quantitative reverse transcription polymerase chain reaction (RT-qPCR) and correlates closely with the clinical results of SeptiCyte LAB, but with a much simpler workflow. Based on the results, the device issues a report with a sepsis probability scale. (see attached algorithm) This new analysis methodology, together with the usual biomarkers, can improve the early diagnosis of sepsis, differentiate between inflamed and septic patients.

The FilmArray® blood culture identification (BCID®) assay is a molecular test approved for direct identification of BSI causing pathogens from positive BC (18). A recently updated version of the panel (BCID2®) comprises improved species identification characteristics and allows for the detection of one expanded-spectrum β-lactamase (ESBL)- and several carbapenemase-encoding genes. The BCID2® Panel tests for 43 targets associated with bloodstream infections, including gram-negative bacteria, gram-positive bacteria, yeast, and 10 antimicrobial resistance genes-all with one test and with results available in about an hour from positive blood culture. In addition, BCID2® Panel menu includes seven additional resistance genes, including carbapenemases, colistin resistance genes and a MREJ assay allows for more speciﬁc MRSA identiﬁcation. A recent study (19) evaluates the clinical performance of the BCID2 assay for species identification in 180 positive blood cultures (BCs). BCID2 results were concordant with the standard of care (SOC) in 159/180 (88.3%) BCs; 68/74 (91.9%) and 71/74 (96.0%) of all samples growing monobacterial, Gram-positive or Gram-negative pathogens, respectively, were identified, in agreement with SOC results.

The usual implementation of the BCID2® is done once the blood culture is positive. However, some preliminary results (20) suggest that the performance of BCID2® in detecting microorganisms very early, may be adequate with only a few hours (6-8h) of blood culture incubation and before the blood culture becomes positive.

Since early diagnosis and early administration of effective antibiotic therapy is of crucial importance to improve patient outcome, the aim of the present study is to develop and evaluate a clinical protocol that combines molecular diagnosis of infection and early determination of microorganisms in blood cultures with only 6-8 hours of incubation before they are found to be positive.

Endpoints

The primary endpoints:

1. - To determine the ability of filmarrays BCID 2® for the early identification of microorganisms in BC with a few hours of incubation and before they have become positive.
2. - To determine the ability of SeptiCyte® for the molecular diagnosis of sepsis in critically ill patients with unclear infectious focus.

The secondary endpoints:

1. - To determine the possible impact of the results on the management of antimicrobial treatment.
2. - To determine if there is an association between common serum biomarkers (PCT, CRP) and positive SeptiCyte® and BCID 2® results.

Main inclusion/exclusion criteria

Inclusion Criteria:

1. - Adults (>16 years old)
2. - At least 2 SIRS criteria
3. - RCP (> 10 mg/dL) or PCT (> 0.5 ng/mL in community or > 1.0ng/mL in nosocomial infection) elevated

3.- Without a clear focus that justifies sepsis 4.- High suspicion of infection that requires starting antimicrobial treatment.

Exclusion criteria:

1. - Failure to obtain the samples within 12 hours after the infection is suspected and antibiotic administration
2. - Previous administration of antimicrobials in the last 24 hours
3. - Documented or evident sepsis focus on ICU admission

Procedures:

MOLECULAR DIAGNOSTIC PROTOCOL AND EARLY DIRECTED TREATMENT (See attached Schedule of Assessments) Once the usual blood samples have been obtained for the determination of PCR, PCT, white blood cell count (WBC) and blood cultures (4 bottles), as well as clinically significant cultures, and if the inclusion criteria are met, the blood cultures (4 bottles) will be sent together with a EDTA tube from those obtained for the usual analysis to the microbiology department where the determination will be carried out with SeptiCyte® and BCID 2® (see attached algorithm).

A) SeptiCyte RAPID® will be performed on all patients at the time of sample receipt in microbiology department. The test result will be stored in the study CRF. This result will not be known to the patient's treating physician.

B) BioFire® FilmArray® blood culture identification panel (BCID 2®) will be performing on the 4 blood culture bottles after 6-8 hours of incubation and especially before it becomes positive. The test result will be stored in the study CRF. This result will not be known to the patient's treating physician. A new BCID 2 determination shall be performed once the blood culture is positive, and the result shall be compared with the one obtained previously with 6-8 hours of incubation.

NOTE: In no case will the information received be used to define behaviours or treatments related to the status of the patient Follow-up Period Patients will be followed up until the event that originated the disorder is considered resolved. Only the first episode of possible sepsis will be considered for each patient.

Patients will be classified as confirmed, probable or possible sepsis according to the definitions from "The International Sepsis Forum Consensus Conference on Definitions of Infection in the Intensive Care Unit. (Calandra T et al. Crit Care Med 2005; 33:1538-1548).

Sample's size calculation According to what was published by Klein Klouwenberg (12), only 25% of patients with suspected of sepsis and who receive antibiotics upon admission to the ICU, are finally classified as having sepsis definitive. The study hopes to be able to identify at least 40% of sepsis in patients with suspected sepsis. Based on this difference and for a power of 90% with an error level of 5%, the number of patients needed to include is 60. Considering a possible loss of 20% of patients (17 patients) the number rises to 100 patients. To ensure the number of patients and the power of the study, it was decided to include a further 20%, making a total of 120 patients.

Data analysis plan:

Qualitative variables will be expressed as percentages, while quantitative variables will be expressed as mean and standard deviation (SD) or median and interquartile range 25-75%. To determine clinical differences between groups with and without BCID 2 and SeptiCyte positives, Chi-square and Fisher tests will be used for categorical variables, and Student's t-test or Mann-Withney U-test for quantitative variables. Multivariate analysis by binary logistic regression will be performed to determine the risk factors associated with the early presence of microorganisms in BCID 2 and for the diagnosis of high risk of sepsis with SeptiCyte.

Finally, an empirical antimicrobial treatment algorithm will be developed for critically ill patients related to the type of microorganisms isolated and the resistance genes evolved.

Limitations The main limitation of the study is the possibility of showing a smaller number of patients with sepsis among the included individuals than the one used to calculate the sample size. This situation could lead to a lack of statistical significance due to the lack of power of the study. To avoid this, it is planned to perform an interim analysis when 70% of the patients are reached. The second limitation is the inclusion of patients at a low rate. Although it has been considered that 6 months of fieldwork will be sufficient, the study could be extended by 4 more months to complete the number of patients.

Ethical considerations The study is being reviewed by the reference Clinical Research and Ethics Committee. Due to its retrospective design and to improve the quality of care, the committee has considered that it is not necessary to request informed consent.

ELIGIBILITY:
Inclusion Criteria:

1. - Age (>15 years old)
2. - At least 2 SIRS criteria
3. - RCP (> 10 mg/dL) or PCT (> 0.5 ng/mL in community or > 1.0ng/mL in nosocomial infection) elevated

3.- Without a clear focus that justifies sepsis 4.- High suspicion of infection that requires starting antimicrobial treatment.

Exclusion Criteria:

1. - Failure to obtain the samples within 12 hours after the infection is suspected and antibiotic administration
2. - Previous administration of antimicrobials in the last 24 hours
3. - Documented or evident sepsis focus on ICU admission

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Critically ill patient who presents with highly suspected sepsis and requires antimicrobial treatment in the next 2-3 hours without evidence of a clear focus responsible for sepsis after an extensive assessment of the patient's condition.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
To determine the ability of filmarryas BCID 2® for the early identification of microorganisms in BC with a few hours of incubation and before they have become positive | Observational period from blood culture collection to 7 days of incubation (period of completion of blood culture incubation when negative results are reported as definitive).
  The number of microorganisms identified by BCID2 after 6-8 hours of incubation with respect to the number of microorganisms identified by blood culture (gold standard).
To determine the ability of SeptiCyte® for the molecular diagnosis of sepsis in critically ill patients with unclear infectious focus. | Observational period from the time of suspected sepsis (defined as the time of blood culture) until resolution of the probable sepsis (usually 7-10 days). Only the first episode of suspected sepsis will be considered for each patient.
  The number of patients classified as having a high, intermediate or no possibility of sepsis with respect to the same classification made on the basis of clinical and laboratory criteria by 3 physicians with expertise in infections at the time of resolution of the suspected sepsis.

SECONDARY OUTCOMES:
To determine the possible impact of the results on the management (optimization) of antimicrobial treatment. | Observational period from the time of suspected sepsis (defined as the time of blood culture) until resolution of the probable sepsis (usually 7-10 days).
  The number of patients in whom antimicrobial treatment was initiated based on clinical criteria with respect to the number of patients requiring antimicrobial treatment (proven sepsis) according to the results of molecular diagnostic techniques (SeptiCyte Rapid and BCID2).

CONTACTS AND LOCATIONS:
Overall Officials: ALEJANDRO RODRIGUEZ, MD,PhD,MSc, Principal Investigator — Hospital Universitari de Tarragona Joan XXIII
Locations (1):
- Alejandro Rodriguez, Tarragona, Spain

REFERENCES:
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Rodriguez A. Sepsis-3: More specific is better? Med Clin (Barc). 2019 Jan 4;152(1):17-18. doi: 10.1016/j.medcli.2018.07.006. Epub 2018 Sep 15. No abstract available. English, Spanish. PMID 30227997
- [Background] Rodriguez A, Martin-Loeches I, Yebenes JC. New definition of sepsis and septic shock: What does it give us? Med Intensiva. 2017 Jan-Feb;41(1):38-40. doi: 10.1016/j.medin.2016.03.008. Epub 2016 May 30. No abstract available. English, Spanish. PMID 27255771
- [Background] Yebenes JC, Ruiz-Rodriguez JC, Ferrer R, Cleries M, Bosch A, Lorencio C, Rodriguez A, Nuvials X, Martin-Loeches I, Artigas A; SOCMIC (Catalonian Critical Care Society) Sepsis Working Group. Epidemiology of sepsis in Catalonia: analysis of incidence and outcomes in a European setting. Ann Intensive Care. 2017 Dec;7(1):19. doi: 10.1186/s13613-017-0241-1. Epub 2017 Feb 20. PMID 28220453
- [Background] Maharaj R, McGuire A, Street A. Association of Annual Intensive Care Unit Sepsis Caseload With Hospital Mortality From Sepsis in the United Kingdom, 2010-2016. JAMA Netw Open. 2021 Jun 1;4(6):e2115305. doi: 10.1001/jamanetworkopen.2021.15305. PMID 34185067
- [Background] Kahn JM, Davis BS, Yabes JG, Chang CH, Chong DH, Hershey TB, Martsolf GR, Angus DC. Association Between State-Mandated Protocolized Sepsis Care and In-hospital Mortality Among Adults With Sepsis. JAMA. 2019 Jul 16;322(3):240-250. doi: 10.1001/jama.2019.9021. PMID 31310298
- [Background] Li AT, Moussa A, Gus E, Paul E, Yii E, Romero L, Lin ZC, Padiglione A, Lo CH, Cleland H, Cheng AC. Biomarkers for the Early Diagnosis of Sepsis in Burns: Systematic Review and Meta-analysis. Ann Surg. 2022 Apr 1;275(4):654-662. doi: 10.1097/SLA.0000000000005198. PMID 35261389
- [Background] Iankova I, Thompson-Leduc P, Kirson NY, Rice B, Hey J, Krause A, Schonfeld SA, DeBrase CR, Bozzette S, Schuetz P. Efficacy and Safety of Procalcitonin Guidance in Patients With Suspected or Confirmed Sepsis: A Systematic Review and Meta-Analysis. Crit Care Med. 2018 May;46(5):691-698. doi: 10.1097/CCM.0000000000002928. PMID 29271844
- [Background] Metlay JP, Waterer GW, Long AC, Anzueto A, Brozek J, Crothers K, Cooley LA, Dean NC, Fine MJ, Flanders SA, Griffin MR, Metersky ML, Musher DM, Restrepo MI, Whitney CG. Diagnosis and Treatment of Adults with Community-acquired Pneumonia. An Official Clinical Practice Guideline of the American Thoracic Society and Infectious Diseases Society of America. Am J Respir Crit Care Med. 2019 Oct 1;200(7):e45-e67. doi: 10.1164/rccm.201908-1581ST. PMID 31573350
- [Background] Kalil AC, Metersky ML, Klompas M, Muscedere J, Sweeney DA, Palmer LB, Napolitano LM, O'Grady NP, Bartlett JG, Carratala J, El Solh AA, Ewig S, Fey PD, File TM Jr, Restrepo MI, Roberts JA, Waterer GW, Cruse P, Knight SL, Brozek JL. Management of Adults With Hospital-acquired and Ventilator-associated Pneumonia: 2016 Clinical Practice Guidelines by the Infectious Diseases Society of America and the American Thoracic Society. Clin Infect Dis. 2016 Sep 1;63(5):e61-e111. doi: 10.1093/cid/ciw353. Epub 2016 Jul 14. PMID 27418577
- [Background] Evans L, Rhodes A, Alhazzani W, Antonelli M, Coopersmith CM, French C, Machado FR, Mcintyre L, Ostermann M, Prescott HC, Schorr C, Simpson S, Wiersinga WJ, Alshamsi F, Angus DC, Arabi Y, Azevedo L, Beale R, Beilman G, Belley-Cote E, Burry L, Cecconi M, Centofanti J, Coz Yataco A, De Waele J, Dellinger RP, Doi K, Du B, Estenssoro E, Ferrer R, Gomersall C, Hodgson C, Moller MH, Iwashyna T, Jacob S, Kleinpell R, Klompas M, Koh Y, Kumar A, Kwizera A, Lobo S, Masur H, McGloughlin S, Mehta S, Mehta Y, Mer M, Nunnally M, Oczkowski S, Osborn T, Papathanassoglou E, Perner A, Puskarich M, Roberts J, Schweickert W, Seckel M, Sevransky J, Sprung CL, Welte T, Zimmerman J, Levy M. Surviving sepsis campaign: international guidelines for management of sepsis and septic shock 2021. Intensive Care Med. 2021 Nov;47(11):1181-1247. doi: 10.1007/s00134-021-06506-y. Epub 2021 Oct 2. No abstract available. PMID 34599691
- [Background] Klein Klouwenberg PM, Cremer OL, van Vught LA, Ong DS, Frencken JF, Schultz MJ, Bonten MJ, van der Poll T. Likelihood of infection in patients with presumed sepsis at the time of intensive care unit admission: a cohort study. Crit Care. 2015 Sep 7;19(1):319. doi: 10.1186/s13054-015-1035-1. PMID 26346055
- [Background] van Vught LA, Wiewel MA, Hoogendijk AJ, Frencken JF, Scicluna BP, Klein Klouwenberg PMC, Zwinderman AH, Lutter R, Horn J, Schultz MJ, Bonten MMJ, Cremer OL, van der Poll T. The Host Response in Patients with Sepsis Developing Intensive Care Unit-acquired Secondary Infections. Am J Respir Crit Care Med. 2017 Aug 15;196(4):458-470. doi: 10.1164/rccm.201606-1225OC. PMID 28107024
- [Background] McHugh L, Seldon TA, Brandon RA, Kirk JT, Rapisarda A, Sutherland AJ, Presneill JJ, Venter DJ, Lipman J, Thomas MR, Klein Klouwenberg PM, van Vught L, Scicluna B, Bonten M, Cremer OL, Schultz MJ, van der Poll T, Yager TD, Brandon RB. A Molecular Host Response Assay to Discriminate Between Sepsis and Infection-Negative Systemic Inflammation in Critically Ill Patients: Discovery and Validation in Independent Cohorts. PLoS Med. 2015 Dec 8;12(12):e1001916. doi: 10.1371/journal.pmed.1001916. eCollection 2015 Dec. PMID 26645559
- [Result] Verboom DM, Koster-Brouwer ME, Varkila MRJ, Bonten MJM, Cremer OL. Profile of the SeptiCyte LAB gene expression assay to diagnose infection in critically ill patients. Expert Rev Mol Diagn. 2019 Feb;19(2):95-108. doi: 10.1080/14737159.2019.1567333. Epub 2019 Feb 5. PMID 30623693
- [Result] Berinson B, Both A, Berneking L, Christner M, Lutgehetmann M, Aepfelbacher M, Rohde H. Usefulness of BioFire FilmArray BCID2 for Blood Culture Processing in Clinical Practice. J Clin Microbiol. 2021 Jul 19;59(8):e0054321. doi: 10.1128/JCM.00543-21. Epub 2021 Jul 19. PMID 33980648
- [Result] Massa-Buck B, Mendoza S, Keiser J, Mohamed MA. Use of Rapid Molecular Polymerase Chain Reaction in Early Detection of Bacteremia in Neonates Prior to Blood Culture Positivity: A Pilot Study. Am J Perinatol. 2024 Apr;41(5):569-574. doi: 10.1055/s-0042-1742743. Epub 2022 Feb 11. PMID 35148542